CLINICAL TRIAL: NCT00748787
Title: Multicenter, Double Blind, Randomized, Controlled With Placebo, to Evaluate the Effect of the Treatment With Plantago Ovata Husk in the Incidence of the Remission of Metabolic Syndrome in Children and Adolescents Between 10 to 16 Years Old.
Brief Title: Trial to Evaluate the Effect of Plantago Ovata Husk in the Remission of Metabolic Syndrome in Children and Adolescents
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was very difficult to fulfill the inclusion criteria, therefore the expected time of inclusion was delayed so much time.
Sponsor: Rottapharm Spain (Industry)
Responsible Party: Anna Anguera, Research Manager
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLAN-EC-PEDIA-01; EudraCT number. 2007-005019-25
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — ispaghula seed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ispaghula husk
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ispaghula husk — 1 sachet of effervescent powder containing 5 gr of product (3.5 g of Ispaghula husk), b.i.d. during 16 weeks. Oral route.
  Other Names: Plantaben
  Arms: 1
Drug: Placebo — 1 sachet of effervescent powder b.i.d. during 16 weeks, oral route.
  Arms: 2

SUMMARY:
The metabolic syndrome represents a constellation of risk factors associated to the abdominal obesity that includes insulin resistance, lipids alterations, high blood pressure etc. Several studies support the hypothesis that the intake of soluble fiber might have a positive effect in the improvement of such of these risk factors.

So that, the aim of this study is to evaluate the efficacy of Ispaghula husk in the remission of metabolic syndrome in children between 10 to 16 years old.

DETAILED DESCRIPTION:
The prevalence of the metabolic syndrome is increasing in the last decade as well in adult people as in children and adolescents. The early diagnosis and treatment measures could be very important in order to reduce the cardiovascular risk in such populations.

Ispaghula husk could be efficacious to reach the remission of the syndrome due to its effects in several important lipidic parameters.

The study will consist in the treatment with Ispaghula husk during 4 months in patients with metabolic syndrome. The main variable is the remission of the metabolic syndrome following the IDF(International Diabetes Federation) criteria specifics for children.

ELIGIBILITY:
Inclusion Criteria:

* Children between 10 to 16 years old with diagnostic criteria of metabolic syndrome following the IDF criteria:

  1. Waist circumference > or equal to percentile 90 according the age.
  2. Presence of 2 or more of following factors: systolic blood pressure > or equal 130 mmHg or diastolic > or equal to 85 mmHg, or treated hypertension
  3. Cholesterol HDL < 1.03 mmol/l or treatment with drugs to increase cHDL
  4. Glucose blood levels > 5.6 mmol/l or type II diabetes diagnosed treated or no.

Exclusion Criteria:

* Loss of body weight > 3kg in the last 2 months
* Waist circumference 10 cm higher of 90 percentile according to the age
* Intake of fiber, aven supplements or phytosterols in the last 2 months
* Glycosylate haemoglobin >7% in the time of inclusion
* Systolic blood pressure > 145 mmHg or Diastolic blood pressure >95 mmHg.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Remission of the metabolic syndrome following the IDF criteria for children, it means, waist circumference lower than 90 percentile of the population according to the age. | 16 weeks

SECONDARY OUTCOMES:
Change in the body weight | 16 weeks
Change in the lipid profile | 16 weeks
Change in the insulin resistance measured by HOMA index | 16 weeks
Change in inflammatory parameters as PCR, IL-6, IL-10, adiponectin | 16 weeks
Changes in blood pressure | 16 weeks
Tolerability of the treatment | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Salas, MD, PhD, Study Chair — Hospital Universitari San Joan de Reus (Tarragona); Luis Peña, MD, PhD, Principal Investigator — Hospital Univer. Materno-Infantil de Canarias ( Las Palmas de Gran Canaria); Margarita Alonso, MD, PhD, Principal Investigator — Hospital Universitario de Valladolid; Sergio Pinillos, MD, Principal Investigator — Hospital Univ. Sant Joan de Déu ( Esplugues de Llobregat, Barcelona); Joan Bel, MD, PhD, Principal Investigator — Hospital Universitari Germans Trias i Pujol ( Badalona); Gloria Bueno, MD, PhD, Principal Investigator — Hosp. Clínico Universitario de Zaragoza; Rosaura Leis, MD, PhD, Principal Investigator — Hospital Clínico Univ. de Santiago de Compostela; Teresa Muñoz, MD, PhD, Principal Investigator — Hospital Univ. del Niño Jesús (Madrid); Albert Feliu, MD PhD, Principal Investigator — Hospital Univ. San Joan de Reus (Tarragona)
Locations (1):
- Hospital Universitari San Joan de Reus, Reus, Tarragona, Spain